CLINICAL TRIAL: NCT01106755
Title: Ground-level Gait Training Combining Body Weight Support and Functional Electrical Stimulation in People Following Chronic Stroke
Brief Title: Effects of Ground Level Gait Training With Body Weight Support (BWS) and Functional Electrical Stimulation (FES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Tania de Fatima Salvini, Universidade Federal de São Carlos
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFSCar-240781
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2008-08

CONDITIONS: Hemiparesis; Stroke
Keywords: kinematic; hemiparesis; gait; Body weight support; Functional electrical stimulation
MeSH Terms: conditions — Paresis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hemiparetic gait (Experimental): gait training on ground level
  Interventions: Device: gait training on ground level using BWS; Device: gait training on ground level using BWS associated to FES

INTERVENTIONS:
Device: gait training on ground level using BWS — An A1-B-A2 system was applied in which A1 and A2 corresponded to gait training on ground level using Body Weight Support (BWS). Each training phase was performed during 45 minutes, three times a week, for six weeks.
Device: gait training on ground level using BWS associated to FES — An A1-B-A2 system was applied in which B corresponded to the training associated to Functional Electrical Stimulation. Each training phase was performed during 45 minutes, three times a week, for six weeks.

SUMMARY:
The aim of this study was to investigate the effects of gait training on ground level, combining BWS and FES in people following chronic stroke.

DETAILED DESCRIPTION:
The body weight support system (BWS) associated to a treadmill as well as to a functional electrical stimulation (FES) of the common peroneal nerve, has been proposed as a strategy for gait training in people following stroke. Moreover, it has also considered that the ground level is the most common locomotion surface, and that there is little information about the effects of gait training, on this kind of surface, in people with hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* Elapsed time since stroke longer than 6 months
* Spasticity classified under level 3 according to the Modified Ashworth Scale
* The ability to walk classified at levels 2, 3 or 4 according to the Functional Ambulation Category

Exclusion Criteria:

* Heart failure, angina pectoris, arrhythmias and other cardiovascular diseases
* Severe lung disease
* Orthopedic disorders
* Cognitive deficits

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
kinematic evaluation | 4 months
  Participants were assessed walking freely at a comfortable self-selected speed before and after each training phase. The analyzed variables were: mean walking speed of locomotion; step length; stride length, speed and duration; initial and final double support duration; single-limb support duration; swing period; range of motion (ROM), maximum and minimum angles of foot, leg, thigh, and trunk segments of both paretic and nonparetic limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Tania F Salvini, PhD, Principal Investigator — Universidade Federal de Sao Carlos (Sao Paulo - Brazil)
Locations (1):
- Universidade Federal de Sao Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Derived] Prado-Medeiros CL, Sousa CO, Souza AS, Soares MR, Barela AM, Salvini TF. Effects of the addition of functional electrical stimulation to ground level gait training with body weight support after chronic stroke. Rev Bras Fisioter. 2011 Nov-Dec;15(6):436-44. doi: 10.1590/s1413-35552011005000030. Epub 2011 Oct 27. PMID 22031271